CLINICAL TRIAL: NCT04601285
Title: A Phase I, Open-label, First-in-human, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of Recombinant Humanized Anti-Trop2 mAb-Tub196 Conjugate in Patients With Advanced Solid Tumors.
Brief Title: A Phase I Study of JS108 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor has adjusted study development plan and terminated this clinical study.
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS108-001-I
Record Dates: First submitted 2020-10-12; First posted 2020-10-23 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental)
  Interventions: Drug: JS108 (recombinant humanized anti-Trop2 mAb-Tub196 conjugate for injection)

INTERVENTIONS:
Drug: JS108 (recombinant humanized anti-Trop2 mAb-Tub196 conjugate for injection) — Dose escalation period: JS108 is administered intravenously every three weeks (Q3W) at the dose corresponding to the enrolled dose cohort.
  Dose expansion period: JS108 is administered intravenously Q3W at the corresponding dose.
  Clinical expansion period: JS108 is administered intravenously Q3W at the recommended dose.

SUMMARY:
This is a phase I, open-label, first-in-human clinical study designed to evaluate the safety, tolerability, PK profile and efficacy of JS108 for patients with advanced solid tumors. This study is divided into 3 periods: dose escalation period, dose expansion period, and clinical expansion period.

ELIGIBILITY:
1. Volunteer to sign an informed consent form.
2. Age of 18-75 years (inclusive), male or female;
3. Expected survival ≥3 months;
4. Histological or cytologically confirmed locally advanced or metastatic solid tumors which progressed on standard of care or with no standard of care available;
5. Toxicity of previous antitumor therapy has recovered to ≤ grade 1 as defined by the NCI-CTCAE v5.0, except alopecia;
6. Subjects dose expansion period and clinical expansion period must have at least one measurable lesion in accordance with RECIST v 1.1;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status score: 0 or 1;
8. Subjects must be able to provide fresh or archived tumor tissue obtained within 1 year prior to inclusion in the study；
9. The organ function level must meet the protocol requirements；
10. Serum pregnancy test confirmed as negative for women of childbearing potential within 7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
First Cycle Dose Limiting Toxicities (DLTs) In Order to Determine the Maximum Tolerated Dose(MTD) | A minimum of 21 days after first infusion of study drug
  Number of participants that experienced dose limiting toxicities(DLTs) at given dose level.
Number of participants with adverse events (AEs) | Through study completion, an average of 1 year
  The adverse events will be evaluated in accordance with CTCAE v5.0. The investigator shall assess the relationship between the events and investigational product.

SECONDARY OUTCOMES:
Maximum observed serum or plasma concentration (Cmax) | Through study completion, an average of 1 year
  One of the pharmacokinetics parameters for JS108
Maximum serum drug time（Tmax） | Through study completion, an average of 1 year
  One of the pharmacokinetics parameters for JS108
Area under the serum or plasma concentration time curve from 0 to infinity (AUC0-inf) | Through study completion, an average of 1 year
  One of the pharmacokinetics parameters for JS108
Volume of distribution at steady state (Vss) | Through study completion, an average of 1 year
  One of the pharmacokinetics parameters for JS108
Terminal phase elimination half life (t½) | Through study completion, an average of 1 year
  One of the pharmacokinetics parameters for JS108
Clearance (CL) | Through study completion, an average of 1 year
  One of the pharmacokinetics parameters for JS108
Anti-drug antibodies (ADA) | Through study completion, an average of 1 year
  To evaluate the immunogenicity of JS108 in patients with advanced solid tumors
Objective Response Rate (ORR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  As determined by the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, which will be complete response (CR) + partial response (PR)
Duration of response (DOR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  DOR is defined as the time from the date of the first documentation of response (confirmed CR or confirmed PR) to the date of the first documentation of PD or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  PFS is defined as the time from the date of randomization to the earlier of the dates of the first documentation of progressive disease or death due to any cause.
Overall Survival (OS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Levels of Trop2 (trophoblast antigen 2) expression in tumor tissue | Through study completion, an average of 1 year
  To investigate any potential correlations of Trop2 levels with responses and toxicity

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality